CLINICAL TRIAL: NCT06398041
Title: Feasibility of Blood Flow Restriction Training in Stroke Patients on a Geriatric Ward
Brief Title: Feasibility BFRT Geriatric Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: S68664
Record Dates: First submitted 2024-04-18; First posted 2024-05-03 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-03

CONDITIONS: Stroke
Keywords: Geriatric patients; Geriatric rehabilitation; Blood Flow Restriction Training; Physiotherapy; Strength training; stroke
MeSH Terms: conditions — Stroke | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Interventional study with the aim to asses the feasibility of this intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Experimental): Patients will undergo 8x a BFRT session and will be asked about their feelings and thoughts using a VAS an 7 points Likert Scale
  Interventions: Other: Blood flow restriction training; Other: Opinions
- Physiotherapists (Other): Physiotherapists involved in the practical application of BFRT will be asked about their thoughts using a 7 point Likert Scale
  Interventions: Other: Opinions

INTERVENTIONS:
Other: Blood flow restriction training — standard physiotherapy 45 minutes per day, 5 day a week (GAPP) + 2 extra sessions of blood flow restriction training
  Arms: Patients
Other: Opinions — Healthcare workers in the geriatric rehabilitation ward and patients will be asked on their opinions on GAPP+Care concerning blood flow restriction training

SUMMARY:
The focus of this interventional study is to assess the feasibility of blood flow restriction training (BFRT) in a geriatric stroke population. Patients will undergo a 4-week program of BFRT additionally to our standard physiotherapy, conducted twice weekly by experienced physiotherapists.

The main goal of the study is to assess its feasibility concerning the safety and tolerance of BFRT from a patients and therapists scope. Furthermore, the investigators want to establish the proportion of eligible individuals & their willingness to undergo BFRT, as well as the time investment.

The feasibility of an effectiveness study and potential sample size will be evaluated aside.

DETAILED DESCRIPTION:
Stroke is often linked to a loss in muscle strength and a decline in functioning during daily life. In the past, several studies have focused on the effects of resistance training on muscle strength in order to restore patients functioning in daily life. For optimal improvements in muscle strength, the use of high loads with few repetitions per set have been recommended, even within the geriatric population. However, the use of high load exercises in a geriatric population can often be challenging, particularly in patients who have suffered a stroke.

To counter this, blood flow restriction training (BFRT) might give some opportunities. BFRT is a relatively new technique for strength training using a cuff to compromise blood flow in combination with low loads. It is a Japanese technique from origin also known as KAATSU and has been proven to be effective in several populations, including a geriatric population.

During this study, patients will undergo 8 sessions of BFRT given by experienced physiotherapists, twice a week during a 4-week program additionally to standard physiotherapy program: the Geriatric Activation Program Pellenberg (GAPP). Each patient will undergo 1 or 2 specific predetermined exercises for the upper or lower limb, based on the individual goals.

The main goal of the study is to assess its feasibility concerning the safety and tolerance of BFRT from a patients and therapists scope. Furthermore, the investigators want to establish the proportion of eligible individuals & their willingness to undergo BFRT, as well as the time investment.

The feasibility of an effectiveness study and potential sample size will be evaluated aside.

ELIGIBILITY:
A. Patients

Inclusion Criteria patients:

* Patients admitted to the geriatric rehabilitation unit
* ≥ 65years old
* Medically stable as determined by the attending physician
* Expecting at least 5 weeks of rehabilitation
* Diagnosis of stroke (haemorrhagic/ischemic)
* medical research council-scores of 2-3/5 for certain muscle groups
* Being able to understand the exercises
* signed informed consent

Exclusion Criteria:

* Skin lesions located at the site of the cuff
* Cognitive impairment making it impossible to understand the exercises
* Severe comorbidities: (Deep Venous Thrombosis; Open wounds or infected wounds; Dialysis; Cancer; Severe High Blood pressure)

B. Healthcare workers:

Inclusion Criteria

* being physiotherapist involved in the practical application of BFRT
* signed informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of eligible individuals and their willingness to undergo BFRT | 1 year
  Number of available patients on the ward and number of eligible patients and number of patients who participate
Prevalence and types of Adverse events | 1 year
  During the entire time frame of the study, all adverse events will be collected and sorted into different categories. Furthermore, the prevalence of this types will be calculated
Rate of attended sessions over the total number of sessions planned | During a time frame of 1 year, this will be calculated during 4weeks/subject
  attended sessions over the total number of sessions planned
Visual Analog Scale for feelings of perceived pain, effort, safety and comfort | During a time frame of 1 year, each subject will be asked to complete a VAS-scale after every trainingssession (8x/subject over a period of 4 weeks)
  Feelings of perceived pain, effort, safety and comfort will be scored after every trainingssession with a visual analog scale
Time investment | 4 weeks/subject
  the time needed to execute the exercises will be divided by the total time (time to prepare the patient, calibrate the cuff pressure and execute the exercises)
Feasibility assessed by the physiotherapist | 1 year
  Feasibility assessed by the physiotherapist using a 7point Likert Scale for an agreement with several statements and will include options: strongly disagree, disagree, somewhat disagree, either agree or disagree, somewhat agree, and agree
Feasibility assessed by the patients | During a time frame of 1 year, this will be calculated during 4weeks/subject
  Feasibility assessed by the patients using a 7point Likert Scale for an agreement with several statements and will include options: strongly disagree, disagree, somewhat disagree, either agree or disagree, somewhat agree, and agree

SECONDARY OUTCOMES:
Muscle Strength 1 | During a time frame of 1 year, each subject will tested at baseline and the day following the last training session (to counteract fatigue) (2 times over 5 weeks/subject)
  The Medical Research Council (MRC) Scale for Muscle Strength, scores ranging from 0 to 5, with higher scores mean a better outcome
Muscle Strength 2 | During a time frame of 1 year, each subject will tested at baseline and the day following the last training session (to counteract fatigue) (2 times over 5 weeks/subject)
  Muscle strength using a handheld dynamometer (MicroFet2), with higher scores mean a better outcome
Active ROM against gravity | During a time frame of 1 year, each subject will tested at baseline and the day following the last training session (to counteract fatigue) (2 times over 5 weeks/subject)
  the active ROM measured with goniometer, with higher scores mean a better outcome
Functional balance | During a time frame of 1 year, each subject will tested at baseline and the day following the last training session (to counteract fatigue) (2 times over 5 weeks/subject)
  Berg Balance Scale (BBS), scores ranging from 0 to 56, with higher scores mean a better outcome
Walking speed | During a time frame of 1 year, each subject will tested at baseline and the day following the last training session (to counteract fatigue) (2 times over 5 weeks/subject)
  10 Meter walking test (10MWT)

CONTACTS AND LOCATIONS:
Overall Officials: Jos Tournoy, MD, Principal Investigator — KU UZ Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, campus Pellenberg, Pellenberg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided